CLINICAL TRIAL: NCT05835271
Title: Exoskeleton Assist to Improve Physical Performance in Patients With Very Severe Chronic Respiratory Disease
Brief Title: Powered Assist Hip Exoskeleton to Improve Ambulation in Severe Lung Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Director, Program in Respiratory Rehabilitation, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XO-Nof1-RCT-RG2023
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lung Disease Chronic
Keywords: Walking; Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: A prospective longitudinal, self-controlled, single-case repeated measures alternating treatment, randomized and counterbalanced cross-over experimental trial design, comparing walking endurance without and with a powered exoskeleton.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exoskeleton assist (Experimental): A powered exoskeleton describes a wearable robot designed around the shape and function of the human body with segments and joints externally coupled to those of the user. The exoskeleton includes a belt frame, sensors that detect a user's desired movements, a computerized controller, motors and actuators, and lightweight batteries.
  Interventions: Device: exoskeleton assist

INTERVENTIONS:
Device: exoskeleton assist — A powered exoskeleton describes a wearable robot designed around the shape and function of the human body with segments and joints externally coupled to those of the user. The exoskeleton includes a rigid outer frame, sensors that detect a user's desired movements, a computerized controller, motors and actuators, and lightweight batteries.
  The exoskeleton is designed to be worn in the community.

SUMMARY:
Chronic respiratory disease (CRD) is among the most prevalent and growing diseases worldwide with disabling consequences. Many with a compromised respiratory system cannot support the metabolic energy demands of walking causing them to walk slowly and stop often. Those with CRD could receive substantial benefit from a powered wearable exoskeleton device that assumes part of the energy of walking. Assisting the legs will lower the metabolic energy demands, and therefore the ventilation required for exercise, thereby allowing them to walk faster and further. Proposed is a series of single-case experiments comparing walking endurance with and without a powered hip exoskeleton assist. The aim of this study is to determine the efficacy of an exoskeleton on walking endurance in ventilatory limited patients with CRD. An exoskeleton could be a novel immediate and long term strategy to augment walking as part of the spectrum of pulmonary rehabilitation and community reintegration.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic respiratory disease
* modified medical research council dyspnoea score (mMRC) ≥ 2

Exclusion Criteria:

* evidence of cardiac rhythm or circulatory compromise
* myocardial infarct within the previous three months
* moderate-severe aortic stenosis
* uncontrolled hypertension
* sustained cardiac arrhythmias
* untreated neoplasia
* lung surgery within the previous three months
* any other predominant co-morbidities or treatments that might influence walk testing
* body size outside of exoskeleton fit specifications
* skin sores or skin breakdown in the area where the device is worn
* a high risk of fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
walking endurance time | an average of 7 tests over 4 weeks
  tolerance (time) of an individualized constant, brisk, walking speed endurance test

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, Principal Investigator — West Park Healthcare Centre
Locations (1):
- Westpark Health Care Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolmage TE, Goldstein RS. Assisting Walking in Patients with Chronic Respiratory Disease Using a Powered Exoskeleton: A Series of N-of-1 Clinical Trials. Ann Am Thorac Soc. 2022 Jul;19(7):1230-1232. doi: 10.1513/AnnalsATS.202201-045RL. No abstract available. PMID 35348445